CLINICAL TRIAL: NCT05501171
Title: Randomized Controlled Trial of a Psychological Mobile Application (App) to Promote Coping for Patients With Acute Myeloid Leukemia (AML)
Brief Title: Psychological Mobile App for Patients With AML
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: the funding agency (blue note therapeutics) pulled out and did not provide funding
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Blue Note Therapeutics (Industry)
Responsible Party: Principal Investigator, El-Jawahri, Areej,M.D., Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 22-257
Record Dates: First submitted 2022-08-12; First posted 2022-08-15 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-07

CONDITIONS: AML; Acute Myeloid Leukemia
Keywords: AML; Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Masking Description: This is a double-blind multi-site randomized efficacy trial of two mobile apps: DreAMLand versus CERENA in 180 patients with AML. Patients will be recruited from 5 sites and randomized in 1:1 fashion, stratified by study site, to DreAMLand versus CERENA. The study investigators and clinicians caring for these patients will be blinded to the study group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DREAMLAND (Experimental): Participants will be recruited from 5 sites and randomized in 1:1 fashion, stratified by study site, to DREAMLAND versus CERENA.
  * Participants will use DREAMLAND and during hospitalization for treatment of AML to learn how to cope most effectively with the diagnosis of AML using an iPad provided by the study team or participant's own iPad.
  * Questionnaires (in-person, over the computer or telephone, or by mail) at predetermined days per protocol days.
  Interventions: Behavioral: DREAMLAND
- CERENA (Active Comparator): Participants will be recruited from 5 sites and randomized in 1:1 fashion, stratified by study site, to DREAMLAND versus CERENA.
  * Participants will use the mobile app CERENA during hospitalization for treatment of AML to learn how to best care for themselves using an iPad provided by the study team or participant's own iPad.
  * Questionnaires (in-person, over the computer or telephone, or by mail) at predetermined days per protocol days.
  Interventions: Behavioral: CERENA

INTERVENTIONS:
Behavioral: DREAMLAND — DREAMLAND is self-administered psychological app for patients with AML that includes four modules, focused on:
  1. Supportive psychotherapy strategies to help patients deal with the initial shock of diagnosis, cope with the loss of independence and abrupt life disruptions, and provide validation and reassurance.
  2. Psychoeducation to manage expectations and enhance preparedness for extended hospitalization and mobilize social support.
  3. Psychosocial skill-building to promote effective coping strategies and facilitate acceptance while living with uncertainty.
  4. Self-care to promote positive health behaviors and enhance patients´ sense of control especially as they transition from the hospital to outpatient care.
  Each module takes 20 minutes to complete. DREAMLAND also includes three optional models that also take 15 minutes to complete.
  Other names BNT200
  Arms: DREAMLAND
Behavioral: CERENA — CERENA is a self-administered physical health app that includes 4 modules focused, focused on:
  1. Education about general wellness.
  2. Nutrition.
  3. Exercise.
  4. Cancer prevention.
  Each module takes 20 minutes to complete. CERENA also includes three optional modules that also take 15 minutes to complete.
  Arms: CERENA

SUMMARY:
This research study is evaluating whether a psychological mobile application (app), is efficacious in reducing anxiety and depression symptoms and improving quality of life for patients diagnosed with acute myeloid leukemia (AML) compared to a physical health promotion app.

DETAILED DESCRIPTION:
Patients with a new diagnosis of AML often confront a sudden and life-threatening diagnosis, requiring an immediate disruption of their life and an urgent 4-6 week hospitalization to initiate intensive chemotherapy. During this hospitalization, they endure substantial physical symptoms due to the side-effects of intensive chemotherapy, which negatively impacts their quality of life. Patients with AML also experience significant psychological distress as they struggle with the abrupt onset of illness, uncertainty regarding their prognosis, physical and social isolation during their hospitalization, and complete loss of independence.

From our prior studies, we learnt that the use of DREAMLAND, a psychological mobile app, was feasible to integrate in the care of patients with AML receiving intensive chemotherapy and has promising efficacy for improving patients' physical and psychological symptoms and their quality of life. In this project, the study doctors want to compare the effectiveness of DREAMLAND versus CERENA in improving the patient experience when diagnosed with AML. CERENA is a mobile app that provides medical information about how to best take care of one´s health. Using this research, the study doctors hope to find out the best way to help patients cope with the diagnosis and treatment for AML.

The study will use questionnaires to measure patient's quality of life, physical symptoms, mood, and the participant sense of control over their situation. Study questionnaires will be completed in the hospital or clinic. The participants will also have the option of completing these questionnaires remotely through a secure web link or through a mailed paper copy.

Blue Note Therapeutics, Inc. is supporting this research study by providing funding. Blue Note Therapeutics is a digital health technology company that focuses on the health needs of patients with a cancer diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients (aged 18 years or older) with a new diagnosis of AML
* Receiving treatment with either a) intensive chemotherapy (7+3) or modification of this regimen on a clinical trial, or b) a similar intensive regimen requiring prolonged 3-6-week hospitalization
* Ability to comprehend and speak English as the mobile apps are only available in English

Exclusion Criteria:

* Patients with a diagnosis of acute promyelocytic leukemia
* Patients with acute or unstable psychiatric or cognitive conditions which the treating clinicians believes prohibits informed consent or compliance with study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2022-10-15 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Anxiety Symptoms | Day 20
  Compare anxiety symptoms between participants receiving DREAMLAND versus CERENA as measured by the Hospital Anxiety and Depression Scale (HADS)-anxiety subscale over 20 days.
  Higher scores on the HADS anxiety subscale (range 0-21) indicate greater anxiety symptoms.

SECONDARY OUTCOMES:
Anxiety Symptoms | Up to Day 90
  Compare anxiety symptoms between participants receiving DREAMLAND versus CERENA as measured by the Hospital Anxiety and Depression Scale (HADS)-anxiety subscale over 90 days.
  Higher scores on the HADS-anxiety subscale (range 0-21) indicate greater anxiety symptoms.
Depression Symptoms | Up to Day 90
  Compare depression symptoms between participants receiving DREAMLAND versus CERENA as measured by the Hospital Anxiety and Depression Scale (HADS)-depression subscale and the Patient Health Questionnaire-9 (PHQ-9) over 90 days.
  Higher scores on the HADS-depression subscale (range 0-21) indicate greater depression symptoms.
  Higher scores on the PHQ-9 (range 0-27) indicate greater depression symptoms.
Quality of Life in Patients with Leukemia | Up to Day 90
  Compare quality of life between participants receiving DREAMLAND versus CERENA as measured by the Functional Assessment of Cancer Therapy-Leukemia (FACT-Leukemia) over 90 days.
  Higher scores on FACT-Leukemia (range 0-176) indicate better quality of life.
Symptom Burden | Up to Day 90
  Compare symptom burden between participants receiving DREAMLAND versus CERENA as measured by the Edmonton Symptom Assessment Scale-Revised (ESAS-R) over 90 days.
  Higher scores on the ESAS-R (range 0-100) indicate worse symptom burden.
Post-Traumatic Stress Disorder (PTSD) Symptoms | Up to Day 90
  Compare PTSD symptoms between participants receiving DREAMLAND versus CERENA as measured by the PTSD Checklist-Civilian Version over 90 days.
  Higher scores on the PTSD Checklist-Civilian Version (range 17-85) indicate greater PTSD symptoms.

OTHER OUTCOMES:
Coping | Up to Day 90
  Compare coping between participants receiving DREAMLAND versus CERENA as measured by the Measure of Current Status - Part A (MOCS-A) over 90 days.
  Higher scores on the MOCS-A (range 0-52) indicate better coping.
Self-efficacy | Up to Day 90
  Compare self-efficacy between participants receiving DREAMLAND versus CERENA as measured by the Cancer Self-Efficacy Scale (CASE) over 90 days.
  Higher scores on the CASE (range 0-170) indicate greater self-efficacy.
Health care utilization | Up to 6 months
  to explore differences in hospitalizations, emergency department visits, and days spent in the hospital between participants receiving DREAMLAND versus CERENA as measured based on data obtained from the Electronic Health Record up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Areej El-Jawahri, MD, Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Duke University, Durham, North Carolina
  - Fred Hutchinson Cancer Research Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation